CLINICAL TRIAL: NCT06772467
Title: The Effect of Reiki and Emotional Release Technique (EFT) on Symptom Burden, Disease Adaptation, Vital Signs and Catheter-Related Pain in Haemodialysis Patients:Randomized Controlled Trial
Brief Title: The Effect of Reiki and EFT on Symptom Burden, Disease Adaptation, Vital Signs and Catheter-Related Pain in HD Patients
Acronym: Reiki-EFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Hakime Aslan, Principal Investigator, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: hanife çelik
Record Dates: First submitted 2024-12-31; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Hemodialysis Patient
Keywords: Reiki; EFT; Hemodialysis; Pain; Symptom
MeSH Terms: conditions — Pain | interventions — Methods; Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reiki group (Experimental): Reiki
  Interventions: Behavioral: Intervention (Reiki)
- EFT group (Experimental): EFT
  Interventions: Behavioral: EFT
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Intervention (Reiki) — Reiki was applied to this group twice a week for 4 weeks by a researcher who had a Reiki application certificate. Reiki sessions were applied to the patients before haemodialysis and the session duration was approximately 35-40 minutes. Reiki is applied to the seven major chakras and many minor chakras in the body. The chakras are located in the centre of the body, on a vertical line, in the front and back of the body. In this study, Reiki was applied to the patients twice a week for 4 weeks. Reiki sessions were performed before haemodialysis and each session lasted approximately 35-40 minutes. The vital signs of the patients were measured and recorded 3 times: before each Reiki session, after the Reiki session, just before the patient entered haemodialysis and after the haemodialysis session. After each session, patients with fistula were asked to mark the level of pain felt during catheter insertion on a visual analogue scale.
  Arms: Reiki group
Behavioral: EFT — Emotional Freedom Technique (EFT) is a method that helps people manage their emotions and disturbing thoughts, helping to reduce their stress and anxiety. EFT is also called tapping.
  EFT sessions were applied to the patients before haemodialysis and the session duration was approximately 35-40 minutes. Patients received 8 sessions of EFT. The vital signs of the patients were measured and recorded 3 times: before each EFT session, after the reiki session, just before the patient entered haemodialysis and after the haemodialysis session. After each session, patients with fistula were asked to mark the level of pain felt during catheter insertion on a visual analogue scale.
  Arms: EFT group

SUMMARY:
Objective: This study was conducted to evaluate the effect of reiki and emotional release technique (EFT) on symptom burden, disease adaptation, vital signs and catheter-related pain in haemodialysis patients.

Method: The study was conducted as a pretest-posttest randomised controlled experimental research model. The study was conducted in two haemodialysis units in Bingöl province between September 2023 and December 2024. The population of the study consisted of all patients receiving treatment in haemodialysis units, and the sample consisted of 96 patients (Reiki group =32, EFT group =32 and control group =32 people) determined by power analysis. "Dialysis symptom index", " Tee end-stage renal failure adjustment scale", "Vital signs follow-up form" and "Visual analogue scale" were used for data collection.

DETAILED DESCRIPTION:
During the research process, 8 sessions of reiki and EFT were applied to the patients in the experimental groups, while the patients in the control group continued to receive routine care practices.

ELIGIBILITY:
Inclusion Criteria:

* To be over 18 years old,
* To agree to participate in the research,
* To be literate,
* To be able to communicate verbally,
* Receiving three sessions of outpatient haemodialysis (HD) treatment per week in the same institution,
* Active use of the fistula,
* No impairment in mental and cognitive functions,
* Receiving HD therapy for at least three months (to be considered a chronic HD programme)

Exclusion Criteria:

* Refusal to participate in research,
* Receiving peritoneal dialysis,
* To have a central venous catheter,
* A psychiatric disorder diagnosed by a psychiatrist,
* To withdraw from the investigation,
* Losing your life in the process of work,
* Change of institution or city,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
The effect of Reiki on dialysis symptoms | 2 month
  Reiki was applied to this group twice a week for 4 weeks by a researcher who had a Reiki application certificate. Reiki sessions were applied to the patients before haemodialysis and the session duration was approximately 35-40 minutes. Pre and post data were obtained 'Dialysis Symptom Index'.
  This index aims to measure the physical and emotional symptoms and their severity experienced by haemodialysis patients in the last seven days. The index consists of 30 items in total and each item describes a different physical or emotional symptom. The symptoms experienced are answered as yes or no, and if the answer is yes, how much this symptom affects the individual is evaluated on a 5-point Likert scale (0: not at all, 4: very much). The score that can be obtained from the index ranges from 0 to 150, and an increase in the score indicates an increase in the severity of the symptom.
The effect of Reiki on compliance to illness | 2 month
  Reiki was applied to this group twice a week for 4 weeks by a researcher who had a Reiki application certificate. Reiki sessions were applied to the patients before haemodialysis and the session duration was approximately 35-40 minutes. Pre and post data were obtained 'End Stage Renal Failure Compliance Scale'.
  This scale consists of four dimensions to assess patients' participation in haemodialysis treatment, medication use, fluid restriction and compliance with dietary recommendations. Each domain has its own scoring system. Scores ranging from 0 to 1200 can be obtained from the scale. An increase in the score indicates an increase in compliance with the disease.
The effect of Reiki on vital sings | 2 month
  Reiki was applied to this group twice a week for 4 weeks by a researcher who had a Reiki application certificate. Reiki sessions were applied to the patients before haemodialysis and the session duration was approximately 35-40 minutes. Pre and post data were obtained "Vital Signs Monitoring Form". The vital signs of the patients were measured and recorded 3 times: before each Reiki session, after the Reiki session, just before the patient entered haemodialysis and after the haemodialysis session.
The effect of Reiki on catheter-related pain | 2 month
  Reiki was applied to this group twice a week for 4 weeks by a researcher who had a Reiki application certificate. Reiki sessions were applied to the patients before haemodialysis and the session duration was approximately 35-40 minutes. Pre and post data were obtained 'Pain Intensity Measurement-Visual Analogue Scale (VAS)' to measure catheter intervention pain. After each session, patients with fistula were asked to mark the level of pain felt during catheter insertion on a visual analogue scale.

SECONDARY OUTCOMES:
The effect of EFT on dialysis symptoms | 2 months
  EFT was applied to this group twice a week for 4 weeks by a researcher who had a EFT application certificate. EFT sessions were applied to the patients before haemodialysis and the session duration was approximately 35-40 minutes. Pre and post data were obtained 'Dialysis Symptom Index'.
  This index aims to measure the physical and emotional symptoms and their severity experienced by haemodialysis patients in the last seven days. The index consists of 30 items in total and each item describes a different physical or emotional symptom. The symptoms experienced are answered as yes or no, and if the answer is yes, how much this symptom affects the individual is evaluated on a 5-point Likert scale (0: not at all, 4: very much). The score that can be obtained from the index ranges from 0 to 150, and an increase in the score indicates an increase in the severity of the symptom.
The effect of EFT on compliance to illness | 2 months
  EFT was applied to this group twice a week for 4 weeks by a researcher who had a EFT application certificate. EFT sessions were applied to the patients before haemodialysis and the session duration was approximately 35-40 minutes.Pre and post data were obtained 'End Stage Renal Failure Compliance Scale'.
  This scale consists of four dimensions to assess patients' participation in haemodialysis treatment, medication use, fluid restriction and compliance with dietary recommendations. Each domain has its own scoring system. Scores ranging from 0 to 1200 can be obtained from the scale. An increase in the score indicates an increase in compliance with the disease.
The effect of EFT on vital sings | 2 months
  EFT was applied to this group twice a week for 4 weeks by a researcher who had a EFT application certificate. EFT sessions were applied to the patients before haemodialysis and the session duration was approximately 35-40 minutes. Pre and post data were obtained "Vital Signs Monitoring Form". The vital signs of the patients were measured and recorded 3 times: before each EFT session, after the EFT session, just before the patient entered haemodialysis and after the haemodialysis session.
The effect of EFT on catheter-related pain | 2 months
  EFT was applied to this group twice a week for 4 weeks by a researcher who had a EFT application certificate. EFT sessions were applied to the patients before haemodialysis and the session duration was approximately 35-40 minutes. Pre and post data were obtained 'Pain Intensity Measurement-Visual Analogue Scale (VAS)' to measure catheter intervention pain. After each session, patients with fistula were asked to mark the level of pain felt during catheter insertion on a visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Hakime Aslan, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aslan H, Pekince H. Nursing students' views on the COVID-19 pandemic and their percieved stress levels. Perspect Psychiatr Care. 2021 Apr;57(2):695-701. doi: 10.1111/ppc.12597. Epub 2020 Aug 17. PMID 32808314